CLINICAL TRIAL: NCT01805193
Title: Validation of Computed Tomography Myocardial Perfusion Imaging Using Quantification of Myocardial Blood Flow by Positron Emission Tomography With 15O-water
Brief Title: Myocardial Blood Flow by 15O Water PET
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 12/SS/0078
Record Dates: First submitted 2013-02-04; First posted 2013-03-06 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; computed tomography myocardial perfusion; positron emission tomography; oxygen 15 labelled water; myocardial perfusion; myocardial blood flow
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected coronary heart disease
  Interventions: Other: Computed tomography myocardial perfusion imaging; Other: Oxygen 15 labelled water positron emission tomography

INTERVENTIONS:
Other: Computed tomography myocardial perfusion imaging
Other: Oxygen 15 labelled water positron emission tomography

SUMMARY:
Coronary heart disease is a very common condition caused by narrowings in the blood vessel supplying the heart. the investigators are studying new tests to diagnose heart disease. In this study the investigators plan to investigate a special scan called a PET/CT (Positron emission tomography/computed tomography) and a new type of CT (Computed tomography) scan to tell us about the flow of blood to the heart muscle.

DETAILED DESCRIPTION:
Participants will undergo PET/CT with oxygen-15 labelled water and computed tomography myocardial perfusion imaging.

ELIGIBILITY:
Inclusion Criteria:

* suspected coronary artery disease

Exclusion Criteria:

* inability or unwillingness to undergo CT or PET imaging
* renal failure (serum creatinine >200 um/L or eGFR <30 ml/min)
* hepatic failure
* allergy to iodinated contrast
* pregnancy
* contraindication to adenosine
* inability to give informed consent
* atrial fibrillation with a fast ventricular rate (>70 beats per minute)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with suspected coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Myocardial blood flow | 1 month
  Myocardial blood flow ( ml/g/min) measured by oxygen-15 water positron emission tomography

SECONDARY OUTCOMES:
Fractional flow reserve | 1 month
  Fractional flow reserve measured during invasive coronary angiography
Myocardial perfusion | 1 month
  Myocardial perfusion measured as hypoperfusion on adenosine computed tomography myocardial perfusion imaging

CONTACTS AND LOCATIONS:
Overall Officials: David Newby, PhD DM, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Imaging Centre, Edinburgh, Scotland, United Kingdom